CLINICAL TRIAL: NCT02708043
Title: The Use of Laryngeal Mask Airway for Adenoidectomies: An Experience of 814 Paediatric Patients
Brief Title: Laryngeal Mask Airway for Adenoidectomies (LMAA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ozlem Ozmete, Medical Doctor, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: KA 15-321
Record Dates: First submitted 2016-02-21; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Adenoidectomy Surgery; Flexible-Laryngeal Mask Airway

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- F-LMA group (Other): LMA were placed to 814 patients for adenoidectomy surgery. Researchers evaluated flexible laryngeal mask airway use during pediatric adenoidectomies in terms of patient safety, comfort, complications and surgeon satisfaction levels.
  Interventions: Other: Flexible-Laryngeal Mask Airway

INTERVENTIONS:
Other: Flexible-Laryngeal Mask Airway

SUMMARY:
The current study retrospectively assesses laryngeal mask airway use during pediatric adenoidectomies in terms of patient safety, comfort, complications and surgeon satisfaction levels.

ELIGIBILITY:
Inclusion Criteria:

* 1-16 years of age
* ASA I-II
* Scheduled for elective adenoidectomy under general anesthesia with F-LMA between June 2012 and November 2015.

Exclusion Criteria:

* Emergency
* Extreme obesity
* Sign of clinical significant infection.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 814 (Actual)
Dates: Start 2012-06; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The incidence of failed LMA (0=failed, 1=good) | 3 year

SECONDARY OUTCOMES:
Surgeon satisfaction level (0=bad, 1=same, 2=good) | 3 year